CLINICAL TRIAL: NCT00178373
Title: Modafinil to Reduce Persistent Fatigue in Patients Following Treatment for Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Principal Investigator, Gary Morrow, Professor, University of Rochester
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U2702
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Cancer; Fatigue; Chemotherapy
Keywords: cancer-related fatigue; chemotherapy; modafinil
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Modafinil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modafinil (Experimental): Modafinil 200 mg taken by mouth once a day. Subjects will take 2 100 mg tablets each morning.
  Interventions: Drug: Modafinil
- placebo (Placebo Comparator): Inactive sugar pill, 2 are taken once a day in the morning
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Modafinil
  Arms: Modafinil
Drug: sugar pill
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the efficacy of modafinil with regard to reducing cancer-related fatigue in cancer patients following chemotherapy or radiation therapy. Secondarily, the effect of modafinil on cognitive dysfunction in the same population will be assessed.

The researchers hypothesize that administering modafinil (PROVIGIL®) to patients experiencing fatigue following completion of cancer treatment will lead to reduction in patient fatigue and prevention of or improvement in patient cognitive dysfunction.

DETAILED DESCRIPTION:
Fatigue is a very common and troublesome side effect experienced in cancer patients before, during and after chemotherapy and radiation treatment. This protocol will increase knowledge about the occurrence and treatment of fatigue that develops during cancer treatments with the rationale that:

1. better control of the fatigue reported by patients during and following cancer treatment is needed,
2. there are few systematic data on the etiology of fatigue following cancer treatment, and
3. there is evidence indicating that chemotherapy is associated with cognitive dysfunction.

Comparisons: In this randomized, placebo-controlled study of cancer patients following their chemotherapy or radiation therapy, we will assess the efficacy of modafinil for relieving cancer-related fatigue by actigraphy and for preventing or improving cognitive dysfunction by computer-generated tasks that have previously been utilized to examine drug-induced changes in performance (CDR Cognitive Assessment). Additional outcome measures will include the Fatigue Symptom Checklist, POMS, Fatigue Severity Scale, sleepiness measured by the Epworth Sleepiness Scale, cytokine blood levels, depression measured by the CES-D, and psychological adjustment to cancer measured by the Mini-MAC.

The primary objective is to:

* compare changes in patient reported fatigue following completion of chemotherapy and/or radiation treatment for cancer in patients who receive open-label modafinil (PROVIGIL®) for 4 weeks

Secondary objectives are to:

* assess the persistence of any effect found with a randomized trial of responders to modafinil or placebo for 4 weeks (responders are those who report at least a 1 point decrease in fatigue as measured by the Brief Fatigue Inventory)
* assess the degree to which modafinil can prevent or reduce cognitive dysfunction following treatment for cancer
* investigate potential relationships among depression, fatigue, cytokines, and cognitive dysfunction

Anticipated results could provide potentially important new information with regard to clinical, theoretical, and methodologic applications; that is, improved pharmacologic and perhaps behavioral control of the debilitating fatigue commonly experienced by patients undergoing treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is longer than one-month post chemotherapy and/or radiation treatment for an initial diagnosis of cancer
* Patient is 18 years of age or older
* Patient is able to swallow medication
* Patient has a Brief Fatigue Inventory (BFI) question #3 "fatigue worst" score of 2 or greater

Exclusion Criteria:

* Patient has ever taken modafinil (PROVIGIL)
* Patient has taken an anticonvulsant for a seizure disorder; has taken any of the following on a regular basis within the past 30 days, a psychostimulant (e.g., amphetamines, methylphenidate [Ritalin], pemoline [Cylert]), or a monoamine oxidase inhibitor (MAOIs)
* Patient has a history of clinically significant cardiac disease, uncontrolled hypertension, alcohol or drug abuse, severe headaches, glaucoma, seizure disorder, narcolepsy, a psychotic disorder, or Tourette's syndrome
* Patient presently taking on a regular basis:

  * an anticoagulant (Coumadin [warfarin], heparin); note that low dose Coumadin (1 mg by mouth daily) given for maintenance of venous access devices is acceptable
  * alpha-interferon or interleukin-2,
  * a corticosteroid (dexamethasone, prednisone, prednisolone)
* Patient has a narrowing (pathological or iatrogenic) or obstruction of the gastrointestinal tract
* Patient is currently pregnant or nursing (if currently using a steroidal contraceptive for fertility control, participant must agree to use a barrier method of contraception during the study and for one full menstrual cycle following the study
* Patient has uncontrolled anemia; receiving treatment for anemia and currently stable is acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2004-05; Primary Completion 2005-12 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
degree to which modafinil can reduce patient fatigue following treatment for cancer | 4 weeks

SECONDARY OUTCOMES:
cytokine blood levels
depression measured by the Center for Epidemiologic Studies-Depression scale (CES-D)
cognitive function measured by the Cognitive Drug Research (CDR) Cognitive Assessment
psychological adjustment to cancer measured by the Mini-Mental Adjustment to Cancer scale (Mini-MAC)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Morrow, Ph.D., M.S., Principal Investigator — University of Rochester, James P. Wilmot Cancer Center, Radiation Oncology Department, Behavioral Medicine Unit, Box 704, 601 Elmwood Avenue, Rochester, NY 14642
Locations (1):
- University of Rochester, James P. Wilmot Cancer Center, Rochester, New York, United States